CLINICAL TRIAL: NCT06080256
Title: Extra Alirocumab in Addition to Statin Therapy in Asymptomatic Intracranial Atherosclerotic Stenosis (EAST-aICAS)----a Pilot Study
Brief Title: Extra Alirocumab in Addition to Statin Therapy in Asymptomatic Intracranial Atherosclerotic Stenosis (EAST-aICAS)
Acronym: EAST-aICAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kezhong Zhang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EAST-aICAS
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Intracranial Atherosclerosis; Atherosclerotic Plaque; Stenosis
Keywords: Alirocumab; asymptomatic; intracranial atherosclerotic stenosis
MeSH Terms: conditions — Intracranial Arteriosclerosis; Plaque, Atherosclerotic; Constriction, Pathologic | interventions — alirocumab; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Patients meeting the enrollment criteria will be randomly assigned to one of the two treatment groups (1:1) and will be followed up for 6 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: investigator-initiated, open-label, blinded endpoint assessment, controlled, randomized pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab added to statin therapy (Experimental): Alirocumab (75 mg every 2 weeks for 6 months) added to statin (Atorvastatin 20-40mg). Anti-platelet aggregation and risk factor management.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Statin therapy (Active Comparator): Atorvastatin 20-40mg. Anti-platelet aggregation and risk factor management in both arms.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Alirocumab — alirocumab (75 mg every 2 weeks)
  Arms: Alirocumab added to statin therapy
Drug: Atorvastatin — Atorvastatin 20-40mg

SUMMARY:
The primary goal of the trial is to investigate whether the lipid lowering strategy using Alirocumab plus statin could cause more changes from baseline in intracranial atherosclerotic plaque and hemodynamic features during 6 months of follow-up, in patients with asymptomatic intracranial artery stenosis.

DETAILED DESCRIPTION:
Intracranial atherosclerosis stenosis (ICAS) is one of the most common causes of stroke worldwide and is particularly prevalent in Asian. It accounts for up to 30-50% of strokes amongst Asian patient cohorts, in contrast to 5-10% of strokes amongst western patient cohorts. The SAMMPRIS established aggressive medical management (Intensive lipid lowering with statin to reach a low-density lipoprotein (LDL)-cholesterol lower than 1.8mmol/L, et al) as a superior choice for symptomatic ICAS compared to the percutaneous transluminal angioplasty and stenting. However, around 15% still had recurrent stroke or death during a median follow-up of 32.4 months in SAMMPRIS study in the aggressive medical management group. On the other hand, in view of the ready availability of MRA or CTA , asymptomatic ICAS (ICAS without causing TIA or stroke) can be found at heath checkup. It would be of great significance to take measures to prevent TIA/stroke in those asymptomatic ICAS.

Alirocumab, a member of proprotein convertase subtilisin-kexin type 9 (PCSK9) inhibitors, is a fully human monoclonal antibody that reduces LDL cholesterol levels by approximately 60%. The ODYSSEY OUTCOMES study showed that Alirocumab reduced the risk of cardiovascular events (e.g. cardiovascular death, myocardial infarction and stroke), in patients with atherosclerotic cardiovascular disease.

This pilot study will recruit 80 patients with asymptomatic intracranial artery stenosis, and directly compare Alirocumab on top of statin with statin therapy in changes of intracranial atherosclerotic plaque and hemodynamic features during 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 years and ≤ 75 years.
2. There is a 50 to 99% stenosis of a major intracranial artery (internal carotid artery [ICA], vertebral artery [VA], basilar artery [BA] and the M1 segment of middle cerebral artery [MCA]). The diagnostic evaluation for ICAS at each site is confirmed by the local investigator, using high resolution MR.
3. There is no TIA or acute ischemic stroke attributed to this ICAS artery; OR, there was an episode of TIA or acute ischemic stroke attributed to this ICAS artery, but this episode occured ≥12 months before randomization.
4. To increase the likelihood that the asymptomatic intracranial stenosis is atherosclerotic, patients aged 30-49 years are required to meet at least one additional criteria (i-vi) below:

   i. insulin dependent diabetes for at least 15 years. ii. at least 2 of the following atherosclerotic risk factors: hypertension (Blood pressure [BP] ≥ 140/90 or on antihypertensive therapy); dyslipidemia (LDL ≥ 130 mg /dl or high density lipoprotein (HDL) < 40 mg/dl or fasting triglycerides ≥150 mg/dl or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event.

   iii. history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease.

   iv. any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic. v. aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography.

   vi. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic.
5. Patient agrees with follow-up visits and is available by phone.
6. Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.

Exclusion Criteria:

1. TIA or acute ischemic stroke attributed to this ICAS artery during the past 12 months before the randomization;
2. Previous treatment of target intracranial lesion with a stent, angioplasty, or other mechanical devices (e.g. mechanical thrombectomy, coil embolization).
3. Plan to perform angioplasty, stenting, coiling, thrombectomy, endarterectomy or aneurysmal coil embolization for target vessels/plaques. In case that patients who receive surgeries during follow-up, they will still be followed up for 6 months.
4. Intracranial tumor (except meningioma) or any intracranial vascular malformation.
5. History of any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural).
6. Intracranial arterial stenosis due to arterial dissection; MoyaMoya disease; any known vasculitic disease; viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebral spinal fluid pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process; reversible cerebral vasoconstriction syndrome (RCVS); suspected recanalized embolus.
7. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%.
8. Use of cholesteryl ester transfer protein (CETP) inhibition treatment, mipomersen, or lomitapide within 12 months prior to randomization. Fenofibrate therapy must be stable for at least 6 weeks prior to final screening at a dose that is appropriate for the duration of the study in the judgment of the investigator. Other fibrate therapy (and derivatives) are prohibited.
9. Prior use of PCSK9 inhibition treatment before this recruitment.
10. Known allergy or contraindication to aspirin, clopidogrel, alirocumab or atorvastatin.
11. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets < 100,000, hematocrit < 30, international normalized ratio (INR) > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), severe liver impairment (aspartate transaminase [AST] or alanine transaminase [ALT] > 3 x normal, cirrhosis), creatine kinase > 5 times the upper limit of normal (ULN) at final screening, severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) < 20mL/min/1.73 square meter at final screening.
12. Major surgery (including open femoral, aortic, cardiac or carotid surgery) within previous 30 days or planned in the 6 months after enrollment.
13. Dementia or psychiatric problem that prevents the patient from relevant evaluation or follow-up reliably.
14. Co-morbid conditions that may limit survival to less than 6 months.
15. Currently breastfeeding, pregnancy, planning to become pregnant and unwilling to use contraception for the duration of this study
16. Enrollment in another study that would conflict with the current study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plaque burden (PB) | This will be assessed at 6 months after recruitment.
  lumen area (LA) is manually contoured on T1-weighted SPACE at the most stenotic site (LAplaque). PB is calculated as (1 - LAplaque/OWAplauqe) × 100%
Degree of stenosis caused by the plaque | This will be assessed at 6 months after recruitment.
  degree of stenosis = (1 - Dplaque/Dreference) × 100%, where Dplaque indicated the diameter of the culprit artery at the most stenotic site, and Dreference was the diameter of the normal artery proximal to the plaque
Plaque enhancement | This will be assessed at 6 months after recruitment.
  grading of plaque enhancement: grade 0 indicated enhancement is similar to or less than that of normal-appearing intracranial arterial walls in the same individual; grade 1, enhancement is greater than that of grade 0 but less than that of the pituitary infundibulum; and grade 2, enhancement is similar to or greater than that of the infundibulum. plaque enhancement ratio (ER): circular region of interest (ROI) was drawn within the plaque on pre-contrast and post-contrast T1-weighted SPACE images, respectively. The mean signal intensity (SI) of plaques were obtained. ER = (SIpost - SIpre)/SIpre ×100%
Remodeling index (RI) of the plaque | This will be assessed at 6 months after recruitment.
  the outer wall area (OWA) is manually contoured on T1-weighted SPACE at the most stenotic site (OWAplaque) and the reference site (OWAreference). RI is calculated as OWAplaque/OWAreference × 100%. Arterial remodeling is categorized as positive if RI > 1.05, intermediate if 0.95 ≤ RI ≤ 1.05, and negative if RI < 0.95;
Presence of T1 hyperintensity in the plaque | This will be assessed at 6 months after recruitment.
  the brightest spot of the plaque with SI >150% of that of the reference vessel wall on pre-contrast T1 image
Plaque distribution: whether it is a concentric plaque or not | This will be assessed at 6 months after recruitment.
  a concentric plaque is defined if the wall involvement was more than 75%, and the minimum wall thickness is higher than 50% of the maximum wall thickness.
Hemodynamic characteristics: Hypoperfusion volume | This will be assessed at 6 months after recruitment.
  dynamic susceptibility contrast-perfusion weighted imaging (DSC-PWI) performed and computed using the singular value decomposition deconvolution method using a commercial software NeuBrainCARE (v1.1.10). Hypoperfusion volume on the ipsilateral side of stroke were automatically calculated by use of time to maximum (Tmax) with time thresholds of > 4 seconds and > 6 seconds, respectively.

SECONDARY OUTCOMES:
Any stroke (ischemic or hemorrhagic) or death during 6 months of follow-up in an intention-to treat analysis. | This will be assessed during 6 months of follow-up.
Changes in LDL-cholesterol levels | This will be assessed during 6 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available to other researchers under the approval of the ethical committee.
Supporting Information: Study Protocol, CSR
Time Frame: the data will be available when summary data are published.

REFERENCES:
- [Background] Holmstedt CA, Turan TN, Chimowitz MI. Atherosclerotic intracranial arterial stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2013 Nov;12(11):1106-14. doi: 10.1016/S1474-4422(13)70195-9. PMID 24135208
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Derived] Chen X, Dai J, Nie P, Gu P, Wang M, Zhang K, Wang Z. Design of the "EAST" strategy in patients with asymptomatic intracranial atherosclerotic stenosis. Clin Neurol Neurosurg. 2024 Oct;245:108507. doi: 10.1016/j.clineuro.2024.108507. Epub 2024 Aug 15. PMID 39182330